CLINICAL TRIAL: NCT01545778
Title: Risk of Shopping Behavior of Tapentadol IR Immediate-Release (IR) Compared to Oxycodone IR Immediate-Release (IR)
Brief Title: Risk of Shopping Behavior of Tapentadol Immediate-Release (IR) Compared to Oxycodone Immediate-Release (IR)
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: VICE PRESIDENT EPIDEMIOLOGY, Janssen R&D US
Other Study IDs: CR100822; RRA-5950 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Substance Abuse Detection
Keywords: Substance abuse detection; Opioids abuse; Tapentadol immediate-release (IR); Oxycodone immediate-release (IR)
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Tapentadol IR
  Interventions: Drug: Tapentadol IR
- Oxycodone IR
  Interventions: Drug: Oxycodone IR

INTERVENTIONS:
Drug: Tapentadol IR — Opioid naive patients exposed to tapentadol IR from July 2009 to December 2010.
  Groups: Tapentadol IR
Drug: Oxycodone IR — Opioid naive patients exposed to Oxycodone IR from July 2009 to December 2010.
  Groups: Oxycodone IR

SUMMARY:
The purpose of this study is to compare the risk of shopping behavior of tapentadol immediate release with the risk of shopping behavior of oxycodone immediate release.

DETAILED DESCRIPTION:
This is a retrospective (a study that looks backward in time, usually using medical records and interviews with patients) matched cohort (designated group followed or traced over a period of time) study using IMS LRx database. This database covers 65% of all retail prescriptions in the United States and includes mail service and specialty pharmacy provider prescriptions independent of the method of payment. The study will include Opioid naive patients exposed to tapentadol immediate release (IR) or oxycodone IR from July 2009 to December 2010. A naive patient is a patient who has not received an opioid of any type in the 3 months before the index date. The index date is the date of the first prescription for tapentadol IR or oxycodone IR after June 30, 2009. Patients will be followed for 1 year from their index dates. Each tapentadol IR-exposed patient will be matched to up to 4 oxycodone IR-exposed patients. Matching will allow to control in the design for potential confounding variables such as time of the exposure, geographic area, specialty of the prescriber, and age. These are variables that have been related with the risk of shopping behavior or abuse.

ELIGIBILITY:
Inclusion Criteria:

* Opioid naive patients (a patient who has not received an opioid of any type in the 3 months before the index date) exposed to tapentadol IR or oxycodone IR from July 2009 to December 2010 [The index date is the date of the first prescription for tapentadol IR or oxycodone IR after June 30, 2009]

Exclusion Criteria:

* Patients with use of any opioid 3 months before the index date
* Patients who within 4 days on or after the index date fill a prescription for a different opioid
* Patients who within 4 days on or after the index date fill a prescription for the same opioid but written by a different prescriber

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Opioid naive patients exposed to tapentadol IR or oxycodone IR from July 2009 to December 2010 who did not fill any other opioid prescription within 4 days on or after the index date. The index date is the date of the first prescription for tapentadol IR or oxycodone IR after June 30, 2009. A naive patient is a patient who has not received an opioid of any type in the 3 months before the index date.
Sampling Method: Non-Probability Sample
Enrollment: 646620 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who developed shopping behavior defined as patients with prescriptions with at least one day of overlap, written by ≥ 2 different prescribers and filled in 3 or more pharmacies | 12 months

SECONDARY OUTCOMES:
Time to first episode of shopping behavior | 12 months
The number of shopping episodes during the year of follow up | 12 months
The type of dispensing in the first episode of shopping event | 12 months
  The type of dispensing in the shopping event will be classified as "Only the indexed opioid" "Indexed opioid was involved", or "Indexed opioid was not involved at all".

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Cepeda MS, Fife D, Vo L, Mastrogiovanni G, Yuan Y. Comparison of opioid doctor shopping for tapentadol and oxycodone: a cohort study. J Pain. 2013 Feb;14(2):158-64. doi: 10.1016/j.jpain.2012.10.012. Epub 2012 Dec 17. PMID 23253635